CLINICAL TRIAL: NCT05762640
Title: Efficacy of Ruxolitinib as First Line Treatment in Primary Haemophagocytic Lymphohistiocytosis (HLH) in Children: a Phase 2, Multicentre, Non-comparative Study
Brief Title: Ruxolitinib as First Line Treatment in Primary Haemophagocytic Lymphohistiocytosis (R-HLH)
Acronym: R-HLH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APHP200023; 2021-006878-23 (EudraCT Number)
Record Dates: First submitted 2023-01-03; First posted 2023-03-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Haemophagocytic Lymphohistiocytosis
Keywords: Haemophagocytic Lymphohistiocytosis; Lymphohistiocytic activation syndrome; Ruxolitinib; Jakavi
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Form: tablets, 50 mg/m2/day in two administrations. Maximum dose is 100 mg/day. Administration in association with Methylprednisolone IV (or Prednisolone PO) starting at 2 mg/kg/day in two administrations.
  Duration of treatment: until D-1 of conditioning for allogeneic HSCT OR 9weeks for patients who are not eligible for HSCT.

SUMMARY:
The purpose of this project is to study the survival of patients until Haematopoietic Stem Cell Transplantation following the use of Ruxolitinib as first-line treatment associated to corticosteroids in primary HLH.

DETAILED DESCRIPTION:
Haemophagocytic lymphohistiocytosis (HLH) is a devastating inflammatory condition caused by uncontrolled proliferation of activated lymphocytes and macrophages secreting an excess of inflammatory cytokines.

Treatment of HLH aims at decreasing inflammation and requires also treatment of the underlying trigger, if any.

The principal goal of the induction therapy is to suppress the life-threatening inflammatory process. Once remission of HLH achieved, patients require allogeneic haematopoietic stem cell transplantation (HSCT), the only curative therapy to date.

Despite significant treatment progress, mortality remains high. The study aims to implement a targeted treatment that is less aggressive than conventional approaches (Etoposide / ATG / Alemtuzumab).

A better understanding of the pathophysiology of primary HLH has opened new avenues for targeted therapy. The central cytokine of the HLH process is IFNγ. IFNγ as well as most cytokines that are elevated in HLH, signal via Janus Kinase (JAK) and Signal Transducer and Activator of Transcription (STAT)-associated receptors. Ruxolitinib, a selective JAK1/2 inhibitor has shown its efficacy in mouse models of HLH, where it significantly reduced disease manifestations and enhanced survival. Notably, Ruxolitinib diminished CD8+ T-cell accumulation and cytokine production, while sparing degranulation and cytotoxicity. Recently, Ruxolitinib has also been used successfully in humans in isolated cases of refractory primary and secondary HLH.

This is a National, phase II, non-comparative and non-randomized, study in France with 9 participating centers. The chosen experimental plan is a Simon's Optimal 2-Step Design.

ELIGIBILITY:
Inclusion Criteria

* Patient aged 0 to 22 years
* Patient with HLH syndrome confirmed by at least one of the two criteria:

  1. Confirmed genetic diagnosis of a condition predisposing to primary HLH (see table 1 and table 2) or abnormal expression of perforin, MUNC13-4, SAP or XIAP in FACS and/or positive family history OR
  2. Presence of at least 5 of the 8 following HLH diagnostic criteria:
* Fever
* Splenomegaly
* Cytopenia (affecting at least two cell lineages)
* Haemoglobin < 9 g/dl (<10 g/dL in neonates)
* Platelets < 100,000/µL
* Absolute neutrophil count (ANC) < 1,000/µL
* Hypertriglyceridemia and/or hypofibrinogenemia
* Fasting triglycerides ≥ 3 mmol/l
* Fibrinogen <1.5 g/L
* Haemophagocytosis found in a histological sample (without evidence of a malignant process or an underlying rheumatic disorder)
* Decreased or absent NK function
* Ferritin ≥ 500 µg/l
* Presence of activated T cells in the immune phenotyping as evidenced by expression of the activation marker DR (superior to the normal value of the laboratory) OR CD25 soluble (sIL-2 receptor) ≥ 2,400 U/mL.
* Patient with no previous specific treatment for HLH syndrome
* For patients of childbearing age : using an effective method of contraception during the trial, and through to 90 days after EOS for male participants and 30 days after EOS for female participants
* Freely given, informed and written consent of legal representative of the participant or consent of the adult participant
* Affiliation to Social Security.

Exclusion Criteria

* Previous treatment with ATG, Alemtuzumab, Etoposide, JAK-inhibitors, rifampicin and/or anti-Interferon gamma antibodies. St. John's Wort, or any other strong CYP3A4 inducers.
* Previous treatment with corticosteroids and/or cyclosporine A for more than 14 days
* Isolated CNS disease.
* Contraindication to receive Ruxolitinib:
* History of hypersensitivity to the active substance or to any of the excipients
* Pregnant or lactating female patient
* Contraindication to receive methylprednisolone or prednisolone
* History of hypersensitivity to the active substance or to any of the excipients
* Any infectious condition with the exception of infections, which are the trigger for lymphohistiocytic activation.
* Patient with acute very severe renal impairment (Creatinine Clearance <15 mL/min/1.73m²) who are NOT receiving dialysis.
* Patient with Grade 4 hepatic failure according to the CTCAE v5.0 of 27 November 2017 (Life-threatening consequences; moderate to severe encephalopathy; coma)
* Past or know active tuberculosis
* Known rheumatologic disorder.
* Known active malignancy.
* Patient who is taking another investigational agent or is enrolled in another treatment protocol.
* Patient who cannot tolerate administration of drugs PO or through NG

Max Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Survival until HSCT | Day 0 until HSCT, up to 8 weeks

SECONDARY OUTCOMES:
Rate of patients achieving a complete response | Day 7, Day 14, Day 21, Day 28, Week 8, and Day-1 of the conditioning for HSCT
  To evaluate the efficacy of Ruxolitinib
Rate of patients achieving a partial response | Day 7, Day 14, Day 21, Day 28, Week 8, and Day-1 of the conditioning for HSCT
  To evaluate the efficacy of Ruxolitinib
Delay to obtain complete response | Day 0 up to Day-1 of the conditioning for HSCT
  To evaluate the efficacy of Ruxolitinib
Delay to obtain partial response | Day 0 up to Day-1 of the conditioning for HSCT
  To evaluate the efficacy of Ruxolitinib
Incidence of HLH reactivation | Day 0 up to Day-1 of the conditioning for HSCT
  HLH reactivation after achieving complete or partial response.
Timing of HLH reactivation | Day 0 up to Day-1 of the conditioning for HSCT
  HLH reactivation after achieving complete or partial response.
Occurrence of a viral infection de novo or worsening of pre-existing viral infection(s) | During Ruxolitinib treatment
  To evaluate treatment tolerance
Occurrence of adverse effects reported in the product information for Ruxolitinib | During Ruxolitinib treatment
  To evaluate treatment tolerance
Concentration of Ruxolitinib in blood | Blood sampling: Day 0, weekly until week 8 of treatment and at Day-8 prior to the conditioning for HSCT
  to evaluate Pharmacokinetics
Concentration of Ruxolitinib in cerebrospinal fluid | Blood sampling: Day 0, weekly until week 8 of treatment and at Day-8 prior to the conditioning for HSCT
  to evaluate Pharmacokinetics
Cytokine profile and gene expression | Day 0, Weekly until week 8 of treatment
  Assess through measurement of IFNγ, TNFα, Interleukin (IL)-6, IL-2, IL-10, IL-18, IL-1b, and CXCL9

CONTACTS AND LOCATIONS:
Overall Officials: Despina MOSHOUS, MD, PhD, Study Chair — Hôpital Necker-Enfants Malades

IPD SHARING:
Plan to Share IPD: No